CLINICAL TRIAL: NCT05721326
Title: Sequential EHR Based Interventions to Increase Genetic Testing for Breast and Ovarian Cancer Predisposition Across Diverse Patient Populations in Gynecology Practices at Penn Medicine
Brief Title: Sequential EHR Based Interventions to Increase Genetic Testing for Breast and Ovarian Cancer Predisposition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 25922; 851980 (Other: IRB)
Record Dates: First submitted 2023-01-30; First posted 2023-02-10 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Genetic Predisposition to Disease; Breast Cancer Female; Ovarian Cancer; Hereditary Breast and Ovarian Cancer; Hereditary Cancer Syndrome; Hereditary Diseases; Gene Mutation-Related Cancer
Keywords: NCCN guidelines; genetic testing; hereditary cancer; breast cancer; ovarian cancer; intervention; sequential intervention; message-based intervention; text message; diverse patient population; genetics; female; digital health technology; germline genetic testing; nudge; EHR based intervention; genetic counseling
MeSH Terms: conditions — Genetic Predisposition to Disease; Ovarian Neoplasms; Hereditary Breast and Ovarian Cancer Syndrome; Neoplastic Syndromes, Hereditary; Genetic Diseases, Inborn; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Eligible patients will be sent a message through the patient portal to encourage genetic counseling and testing. If the patient does not respond, they will be sent a text message. Should there be no response, the patient's clinician will receive a nudge
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequential Communications (Experimental): This sequential arm contains three types of communication to be employed following non-response to the previous type. The initial communication will be a direct message to the patient via the MyPennMedicine. The subsequent message will be sent as a text via the Way To Health app(lication). The final communication will be a nudge to the patient's physician which will send upon opening the patient's chart and will remain as a flag thereafter.
  Interventions: Other: Sequential EHR Communications

INTERVENTIONS:
Other: Sequential EHR Communications — The intervention includes 3 message types: an EHR message, followed by a text message, followed by physician nudge. Each subsequent type will be activated if the previous type does not yield a response.

SUMMARY:
The goal of this sequential study design is to increase genetic testing in those meeting national clinical guidelines. The main question it aims to answer is: which intervention is most effective in uptake of genetic testing for the target population? Participants will receive genetic testing and counseling that may initiate life-saving screenings.

DETAILED DESCRIPTION:
Germline genetic testing is recommended by the National Cancer Center Network (NCCN) for individuals with a personal history of ovarian cancer, young-onset (<50 years) breast cancer, and a family history of ovarian cancer or male breast cancer, among others. Recent publications demonstrate that the uptake of genetic testing is under-utilized, overall, and rates are consistently lower in minority populations. EHR-based algorithms will be used to identify patients of two Penn Medicine Ob/Gyn practices for whom genetic testing is recommended based on NCCN guidelines and to test pragmatic methods using messages delivered to patients or clinicians to encourage testing. The ACC Electronic Phenotyping Core developed the algorithms based on cancer registry data along with family history fields and this study will develop and test messages directed at patients and clinicians to encourage testing. The aims are:

1. Identification of at-risk populations through electronic health record (EHR) searches followed by patient nudges (MPM and then Way To Health) to increase the uptake of genetic counseling referral and testing in patients at gynecology practices at Dickens Center and Penn Medicine Radnor.
2. In patients who have not responded to patient nudges (Aim 1), test a provider nudge to increase the uptake of genetic counseling referral and testing in gynecology practices at Dickens Center and Penn Medicine Radnor (Aim 2).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with serous ovarian cancer diagnosed more than two years prior to study contact
2. Patients with breast cancer diagnosed at <50 years of age more than two years prior to study contact
3. Patients with triple negative breast cancer diagnosed more than two years prior to study contact
4. Unaffected individuals reporting a family history of ovarian cancer
5. Unaffected individuals reporting a family history of male breast cancer
6. Unaffected individuals reporting a family history of breast cancer <50 years

Exclusion Criteria:

1. Patients who have previously received genetic counseling and/or testing

Ages: 25 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1330 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Number of Genetic Counseling Appointments Completed Following MPM Delivery | Within six months of MPM delivery
  Scheduling and completion of genetic counseling appointments will be monitored through EHR. MPM stands for MyPennMedicine message which will be sent directly to the patient through the medical record.
Number of Genetic Counseling Appointments Completed Following Provider Nudge | Within six months of provider nudge
  Scheduling and completion of genetic counseling appointments will be monitored through EHR. The provider nudge will be delivered as a Best Practice Alert (BPA) upon opening the patient's chart.

SECONDARY OUTCOMES:
Open Rate of MPM | Within one month of receiving MPM
  The proportion of eligible participants who open the invitation to receive genetic counseling and testing compared to the total amount of eligible participants sent an MPM.
Response Rate of Way To Health text | Within one month of receiving text
  The proportion of eligible participants who respond to a text message invitation to receive genetic counseling and testing compared to the total amount of eligible participants sent a Way To Health (WTH) text.

OTHER OUTCOMES:
Number of Signed Referrals | Within one month of receiving referral
  The total number of referrals signed by the patient's Ob/Gyn provider for genetic counseling and testing.

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Srivastava SK, Ahmad A, Miree O, Patel GK, Singh S, Rocconi RP, Singh AP. Racial health disparities in ovarian cancer: not just black and white. J Ovarian Res. 2017 Sep 21;10(1):58. doi: 10.1186/s13048-017-0355-y. PMID 28931403
- [Background] Menon U, Gentry-Maharaj A, Burnell M, Singh N, Ryan A, Karpinskyj C, Carlino G, Taylor J, Massingham SK, Raikou M, Kalsi JK, Woolas R, Manchanda R, Arora R, Casey L, Dawnay A, Dobbs S, Leeson S, Mould T, Seif MW, Sharma A, Williamson K, Liu Y, Fallowfield L, McGuire AJ, Campbell S, Skates SJ, Jacobs IJ, Parmar M. Ovarian cancer population screening and mortality after long-term follow-up in the UK Collaborative Trial of Ovarian Cancer Screening (UKCTOCS): a randomised controlled trial. Lancet. 2021 Jun 5;397(10290):2182-2193. doi: 10.1016/S0140-6736(21)00731-5. Epub 2021 May 12. PMID 33991479
- [Background] Reid S, Cadiz S, Pal T. Disparities in Genetic Testing and Care among Black women with Hereditary Breast Cancer. Curr Breast Cancer Rep. 2020 Sep;12(3):125-131. doi: 10.1007/s12609-020-00364-1. Epub 2020 May 19. PMID 33603954
- [Background] Jatoi I, Sung H, Jemal A. The Emergence of the Racial Disparity in U.S. Breast-Cancer Mortality. N Engl J Med. 2022 Jun 23;386(25):2349-2352. doi: 10.1056/NEJMp2200244. Epub 2022 Jun 18. No abstract available. PMID 35713541
- [Background] Domchek SM, Robson ME. Update on Genetic Testing in Gynecologic Cancer. J Clin Oncol. 2019 Sep 20;37(27):2501-2509. doi: 10.1200/JCO.19.00363. Epub 2019 Aug 12. No abstract available. PMID 31403865
- [Background] Daly MB, Pal T, Berry MP, Buys SS, Dickson P, Domchek SM, Elkhanany A, Friedman S, Goggins M, Hutton ML; CGC; Karlan BY, Khan S, Klein C, Kohlmann W; CGC; Kurian AW, Laronga C, Litton JK, Mak JS; LCGC; Menendez CS, Merajver SD, Norquist BS, Offit K, Pederson HJ, Reiser G; CGC; Senter-Jamieson L; CGC; Shannon KM, Shatsky R, Visvanathan K, Weitzel JN, Wick MJ, Wisinski KB, Yurgelun MB, Darlow SD, Dwyer MA. Genetic/Familial High-Risk Assessment: Breast, Ovarian, and Pancreatic, Version 2.2021, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2021 Jan 6;19(1):77-102. doi: 10.6004/jnccn.2021.0001. PMID 33406487
- [Background] Smith-Uffen M, Bartley N, Davies G, Best M. Motivations and barriers to pursue cancer genomic testing: A systematic review. Patient Educ Couns. 2021 Jun;104(6):1325-1334. doi: 10.1016/j.pec.2020.12.024. Epub 2020 Dec 25. PMID 33390305
- [Background] Kurian AW, Ward KC, Howlader N, Deapen D, Hamilton AS, Mariotto A, Miller D, Penberthy LS, Katz SJ. Genetic Testing and Results in a Population-Based Cohort of Breast Cancer Patients and Ovarian Cancer Patients. J Clin Oncol. 2019 May 20;37(15):1305-1315. doi: 10.1200/JCO.18.01854. Epub 2019 Apr 9. PMID 30964716
- [Background] McBride CM, Pathak S, Johnson CE, Alberg AJ, Bandera EV, Barnholtz-Sloan JS, Bondy ML, Cote ML, Moorman PG, Peres LC, Peters ES, Schwartz AG, Terry PD, Schildkraut JM. Psychosocial factors associated with genetic testing status among African American women with ovarian cancer: Results from the African American Cancer Epidemiology Study. Cancer. 2022 Mar 15;128(6):1252-1259. doi: 10.1002/cncr.34053. Epub 2021 Dec 9. PMID 34882782
- [Background] Hamilton JG, Symecko H, Spielman K, Breen K, Mueller R, Catchings A, Trottier M, Salo-Mullen EE, Shah I, Arutyunova A, Batson M, Gebert R, Pundock S, Schofield E, Offit K, Stadler ZK, Cadoo K, Carlo MI, Narayan V, Reiss KA, Robson ME, Domchek SM. Uptake and acceptability of a mainstreaming model of hereditary cancer multigene panel testing among patients with ovarian, pancreatic, and prostate cancer. Genet Med. 2021 Nov;23(11):2105-2113. doi: 10.1038/s41436-021-01262-2. Epub 2021 Jul 13. PMID 34257420
- [Background] Lau-Min KS, Guerra CE, Nathanson KL, Bekelman JE. From Race-Based to Precision Oncology: Leveraging Behavioral Economics and the Electronic Health Record to Advance Health Equity in Cancer Care. JCO Precis Oncol. 2021 Feb 17;5:PO.20.00418. doi: 10.1200/PO.20.00418. eCollection 2021. No abstract available. PMID 34250405
- [Background] Kukafka R, Pan S, Silverman T, Zhang T, Chung WK, Terry MB, Fleck E, Younge RG, Trivedi MS, McGuinness JE, He T, Dimond J, Crew KD. Patient and Clinician Decision Support to Increase Genetic Counseling for Hereditary Breast and Ovarian Cancer Syndrome in Primary Care: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2022 Jul 1;5(7):e2222092. doi: 10.1001/jamanetworkopen.2022.22092. PMID 35849397
- [Derived] Symecko H, Schnoll R, Beidas RS, Bekelman JE, Blumenthal D, Bauer AM, Gabriel P, Boisseau L, Doucette A, Powers J, Cappadocia J, McKenna DB, Richardville R, Cuff L, Offer R, Clement EG, Buttenheim AM, Asch DA, Rendle KA, Shelton RC, Fayanju OM, Wileyto EP, Plag M, Ware S, Shulman LN, Nathanson KL, Domchek SM. Protocol to evaluate sequential electronic health record-based strategies to increase genetic testing for breast and ovarian cancer risk across diverse patient populations in gynecology practices. Implement Sci. 2023 Nov 6;18(1):57. doi: 10.1186/s13012-023-01308-w. PMID 37932730